CLINICAL TRIAL: NCT02889497
Title: Safety, Three Batches Consistency and Immunity Duration of the Post-marketing Inactivated Enterovirus Type 71 (EV71) Vaccine in Children Aged 6-71 Months
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cycdc2016-6
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Hand Foot and Mouth Disease
Keywords: vaccine; safety; immunogenicity
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 300 subjects receive the first batch vaccine (Experimental): 300 subjects will be randomly received the first batch vaccine
  Interventions: Biological: the first batch vaccine
- 300 subjects receive the second batch vaccine (Experimental): 300 subjects will be randomly received the second batch vaccine
  Interventions: Biological: the second batch vaccine
- 300 subjects receive the third batch vaccine (Experimental): 300 subjects will be randomly received the third batch vaccine
  Interventions: Biological: the third batch vaccine

INTERVENTIONS:
Biological: the first batch vaccine
  Arms: 300 subjects receive the first batch vaccine
Biological: the second batch vaccine
  Arms: 300 subjects receive the second batch vaccine
Biological: the third batch vaccine
  Arms: 300 subjects receive the third batch vaccine

SUMMARY:
This study evaluates the safety,three batches consistency and immunity duration of the post-marketing inactivated Enterovirus Type 71 (EV71) vaccine in children aged 6-71 months.This study has two groups:safety observation group and immunogenicity observation group.20000 subjects will receive 2 doses vaccines and be observed for safety among 2 epidemic cycles of HFMD.In the immunogenicity observation group, 900 subjects will be randomly received 3 batches vaccines(2 doses),and blood sampled at days 0 and 56.

ELIGIBILITY:
Inclusion Criteria:

* 8 Months to 71 Months (Healthy Children or Infants)；
* Providing the subjects' legal identity certificate (birth certificate , residence booklet or ID card) and vaccination certificate, legal guardians can provide legal identity proof (resident booklet or ID card) so that the doctor can determine the subject identity to complete recruitment program；
* The subjects' guardians are able to understand and sign the informed consent voluntary. Guardians have the ability to use the thermometer ,dividing ruler and can fill out the Diary card ,follow-up card according to requirements；
* Persist for a 24 months visit.If doubtful HFMD case happen，the subject's guardian should send the subject to the medical institutions at above the county level and report this case to the investigator.The subjects who participate immunogenicity observation group can receive sample collection including blood，throat swab or anal awab according to program requirements.

Exclusion Criteria:

* Exclusion Criteria for the first dose:

  * Subject with clinical diagnosis or suspect HFMD（Especially the history of herpangina）；
  * Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine；
  * History of seizures,convulsions or twitching ;Family history of progressive neurological disease；
  * Autoimmune disease or immunologic deficiency.Any prior administration of immunodepressant in last 6month；
  * History of asthma，thyroid ablation，angioneurotic edema, diabetes mellitus or malignant tumour；
  * Alienia，functional asplenia，or any condition that cause asplenia or splenectomy；
  * Diagnosed coagulation abnormalities (such as clotting factor deficiency, coagulation disorders, platelet disorder) or significant bruising or blood clotting disorder；
  * Any acute disease or chronic disease attack in last 7 days；
  * Any prior administration of blood products in last 3 month；
  * Any prior administration of attenuated live vaccine in last 15 days , subunit or inactivated vaccines in last 7 days；
  * Fever before vaccination, axillary temperature ﹥37.0℃；
  * Attend Other vaccine or drug clinical trials concurrent in 6 months；
  * Any condition that in the opinion of the investigator。
* Exclusion Criteria for the second dose:

  * Any exclusion criteria for the first dose happens after been enrolled；
  * Newly HFMD diagnosed patients after been enrolled；
  * Any condition that in the opinion of the investigator or ethics committee think should be eliminated.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20900 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Rate of Adverse reactions of Post-marketing Inactivated Enterovirus Type 71 (EV71) Vaccine in Children Aged 6-71 Months. | 24 months
  Adverse reactions associated with vaccine will be observed in Children Aged 6-71 Months after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy.
Evaluate the seroconversion rate of EV71 antibodies in serum after vaccination. | 56 days
  The seroconversion rate of EV71 antibodies will be evaluated in serum at days 0 and 56.